CLINICAL TRIAL: NCT03208920
Title: Omega EVAR: Use of Fish Oil to Reduce Inflammation During Endovascular Abdominal Aortic Repair.
Brief Title: Use of Fish Oil to Reduce Inflammation During Endovascular Abdominal Aortic Repair
Acronym: Omega-EVAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-16505
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: PAD; Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pro-Omega (Experimental): High-dose, short-duration dietary omega-3 fatty acids supplementation; 4400 mg/day x 6 months (Nordic Naturals, Watsonville, CA, USA)
  Interventions: Dietary Supplement: Pro-Omega
- Placebo (Placebo Comparator): Pro-Omega Placebo soybean capsules (Nordic Naturals, Watsonville, CA, USA); 4400mg/day x 6 months
  Interventions: Other: ProOmega Placebo

INTERVENTIONS:
Dietary Supplement: Pro-Omega — Pro-Omega (Nordic Naturals, Watsonville, CA, USA). Each Pro-Omega capsule is 550 mg. Must take 4400 mg/day x 6 months.
  Arms: Pro-Omega
Other: ProOmega Placebo — Placebo Comparator: soybean (Nordic Naturals, Watsonville, CA, USA). Each soybean capsule is 550 mg. Must take 4400 mg/day x 6 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if high-dose PUFA supplementation in patients undergoing EVAR for infra-renal AAA reduces the peri-operative inflammation.

DETAILED DESCRIPTION:
In this 2:1 double-blind, randomized, placebo controlled trial, subjects will be given an active drug of n-3 polyunsaturated fatty acids (PUFAs) or a placebo soybean oil for about two weeks prior to an endovascular abdominal aortic repair (EVAR) and subsequently six months after the procedure.

An EVAR is known to produce a systemic inflammatory response with an increased risk of prolonged hospitalization and complicated post-operative recovery with cardiac events, renal and pulmonary dysfunction, and multiple organ failure. The study proposed here has the potential to provide valuable insight on the role of nutritional intervention to improve outcomes related to surgical revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing EVAR for infra-renal AAA and/or iliac artery aneurysm

Exclusion Criteria:

* Age < 40 or > 90 years
* On dual antiplatelet therapy or anticoagulation
* Evidence of active infection
* Diagnosed hypercoagulable state
* Non-atherosclerotic/aneurysmal disease as indication for procedure
* Chronic liver disease or myopathy
* End-stage renal disease (CKD 5)
* Poorly controlled diabetes (HbA1C > 8%)
* Recent other major surgery or illness within 6 weeks
* Use of immunosuppressive medication or extant chronic inflammatory disorders
* History of organ transplantation
* Pregnancy or plans to become pregnant
* Condition in which patient life expectancy is less than one year
* Known allergy to fish or fish products
* Presence of symptomatic or ruptured AAA

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Highly Sensitive C-Reactive Protein | 6 months
  Blunting of the peri-PVI inflammatory response as measured by the area under the curve (AUC) of the inflammatory biomarker high sensitivity C reactive protein (CRP)

SECONDARY OUTCOMES:
Systemic Inflammatory Markers | 6 months
  Reduce circulating pro-inflammatory markers (PIMs) and increase pro-resolution mediators (PRMs) assayed using targeted metabolo-lipidomics, increase PRM production within peripheral circulating monocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Warren Gasper, M.D, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco Veteran Affairs Medical Center, San Francisco, California, United States

REFERENCES:
- [Background] Galle C, De Maertelaer V, Motte S, Zhou L, Stordeur P, Delville JP, Li R, Ferreira J, Goldman M, Capel P, Wautrecht JC, Pradier O, Dereume JP. Early inflammatory response after elective abdominal aortic aneurysm repair: a comparison between endovascular procedure and conventional surgery. J Vasc Surg. 2000 Aug;32(2):234-46. doi: 10.1067/mva.2000.107562. PMID 10917982
- [Background] Serhan CN, Brain SD, Buckley CD, Gilroy DW, Haslett C, O'Neill LA, Perretti M, Rossi AG, Wallace JL. Resolution of inflammation: state of the art, definitions and terms. FASEB J. 2007 Feb;21(2):325-32. doi: 10.1096/fj.06-7227rev. PMID 17267386
- [Background] Serhan CN, Chiang N, Van Dyke TE. Resolving inflammation: dual anti-inflammatory and pro-resolution lipid mediators. Nat Rev Immunol. 2008 May;8(5):349-61. doi: 10.1038/nri2294. PMID 18437155
- [Background] Serhan CN, Hong S, Gronert K, Colgan SP, Devchand PR, Mirick G, Moussignac RL. Resolvins: a family of bioactive products of omega-3 fatty acid transformation circuits initiated by aspirin treatment that counter proinflammation signals. J Exp Med. 2002 Oct 21;196(8):1025-37. doi: 10.1084/jem.20020760. PMID 12391014
- [Background] Spite M, Serhan CN. Novel lipid mediators promote resolution of acute inflammation: impact of aspirin and statins. Circ Res. 2010 Nov 12;107(10):1170-84. doi: 10.1161/CIRCRESAHA.110.223883. PMID 21071715
- [Background] Serhan CN. Resolution phase of inflammation: novel endogenous anti-inflammatory and proresolving lipid mediators and pathways. Annu Rev Immunol. 2007;25:101-37. doi: 10.1146/annurev.immunol.25.022106.141647. PMID 17090225
- [Background] Serhan CN, Yang R, Martinod K, Kasuga K, Pillai PS, Porter TF, Oh SF, Spite M. Maresins: novel macrophage mediators with potent antiinflammatory and proresolving actions. J Exp Med. 2009 Jan 16;206(1):15-23. doi: 10.1084/jem.20081880. Epub 2008 Dec 22. PMID 19103881
- [Background] Ho KJ, Spite M, Owens CD, Lancero H, Kroemer AH, Pande R, Creager MA, Serhan CN, Conte MS. Aspirin-triggered lipoxin and resolvin E1 modulate vascular smooth muscle phenotype and correlate with peripheral atherosclerosis. Am J Pathol. 2010 Oct;177(4):2116-23. doi: 10.2353/ajpath.2010.091082. Epub 2010 Aug 13. PMID 20709806
- [Background] Grenon SM, Conte MS, Nosova E, Alley H, Chong K, Harris WS, Vittinghoff E, Owens CD. Association between n-3 polyunsaturated fatty acid content of red blood cells and inflammatory biomarkers in patients with peripheral artery disease. J Vasc Surg. 2013 Nov;58(5):1283-90. doi: 10.1016/j.jvs.2013.05.024. Epub 2013 Jul 2. PMID 23830313
- [Background] Wang JH, Eguchi K, Matsumoto S, Fujiu K, Komuro I, Nagai R, Manabe I. The omega-3 polyunsaturated fatty acid, eicosapentaenoic acid, attenuates abdominal aortic aneurysm development via suppression of tissue remodeling. PLoS One. 2014 May 5;9(5):e96286. doi: 10.1371/journal.pone.0096286. eCollection 2014. PMID 24798452
- [Background] Velazquez OC, Carpenter JP, Baum RA, Barker CF, Golden M, Criado F, Pyeron A, Fairman RM. Perigraft air, fever, and leukocytosis after endovascular repair of abdominal aortic aneurysms. Am J Surg. 1999 Sep;178(3):185-9. doi: 10.1016/s0002-9610(99)00144-0. PMID 10527435
- [Background] Storck M, Scharrer-Pamler R, Kapfer X, Gallmeier U, Gorich J, Sunder-Plassmann L, Bruckner U, Mickley V. Does a postimplantation syndrome following endovascular treatment of aortic aneurysms exist? Vasc Surg. 2001 Jan-Feb;35(1):23-9. doi: 10.1177/153857440103500105. PMID 11668365
- [Background] Rizas KD, Ippagunta N, Tilson MD 3rd. Immune cells and molecular mediators in the pathogenesis of the abdominal aortic aneurysm. Cardiol Rev. 2009 Sep-Oct;17(5):201-10. doi: 10.1097/CRD.0b013e3181b04698. PMID 19690470
- [Background] Lindeman JH, Abdul-Hussien H, Schaapherder AF, Van Bockel JH, Von der Thusen JH, Roelen DL, Kleemann R. Enhanced expression and activation of pro-inflammatory transcription factors distinguish aneurysmal from atherosclerotic aorta: IL-6- and IL-8-dominated inflammatory responses prevail in the human aneurysm. Clin Sci (Lond). 2008 Jun;114(11):687-97. doi: 10.1042/CS20070352. PMID 18078385
- [Background] Zimmer S, Heiss MM, Schardey HM, Weilbach C, Faist E, Lauterjung L. [Inflammatory syndrome after endovascular implantation of an aortic stent--a comparative study]. Langenbecks Arch Chir Suppl Kongressbd. 1998;115(Suppl I):13-7. German. PMID 14518202
- [Background] Boyle JR, Goodall S, Thompson JP, Bell PR, Thompson MM. Endovascular AAA repair attenuates the inflammatory and renal responses associated with conventional surgery. J Endovasc Ther. 2000 Oct;7(5):359-71. doi: 10.1177/152660280000700503. PMID 11032254
- [Background] Chang CK, Chuter TA, Niemann CU, Shlipak MG, Cohen MJ, Reilly LM, Hiramoto JS. Systemic inflammation, coagulopathy, and acute renal insufficiency following endovascular thoracoabdominal aortic aneurysm repair. J Vasc Surg. 2009 May;49(5):1140-6. doi: 10.1016/j.jvs.2008.11.102. PMID 19394543
- [Background] Moulakakis KG, Alepaki M, Sfyroeras GS, Antonopoulos CN, Giannakopoulos TG, Kakisis J, Karakitsos P, Liapis CD. The impact of endograft type on inflammatory response after endovascular treatment of abdominal aortic aneurysm. J Vasc Surg. 2013 Mar;57(3):668-77. doi: 10.1016/j.jvs.2012.09.034. Epub 2013 Jan 11. PMID 23317524
- [Background] Morikage N, Esato K, Zenpo N, Fujioka K, Takenaka H. Is endovascular treatment of abdominal aortic aneurysms less invasive regarding the biological responses? Surg Today. 2000;30(2):142-6. doi: 10.1007/PL00010062. PMID 10664337
- [Background] Swartbol P, Truedsson L, Norgren L. Adverse reactions during endovascular treatment of aortic aneurysms may be triggered by interleukin 6 release from the thrombotic content. J Vasc Surg. 1998 Oct;28(4):664-8. doi: 10.1016/s0741-5214(98)70092-8. PMID 9786262
- [Background] Gerasimidis T, Sfyroeras G, Trellopoulos G, Skoura L, Papazoglou K, Konstantinidis K, Karamanos D, Filaktou A, Parapanisiou E. Impact of endograft material on the inflammatory response after elective endovascular abdominal aortic aneurysm repair. Angiology. 2005 Nov-Dec;56(6):743-53. doi: 10.1177/000331970505600612. PMID 16327951
- [Background] Serhan CN, Savill J. Resolution of inflammation: the beginning programs the end. Nat Immunol. 2005 Dec;6(12):1191-7. doi: 10.1038/ni1276. PMID 16369558
- [Background] Bannenberg GL, Chiang N, Ariel A, Arita M, Tjonahen E, Gotlinger KH, Hong S, Serhan CN. Molecular circuits of resolution: formation and actions of resolvins and protectins. J Immunol. 2005 Apr 1;174(7):4345-55. doi: 10.4049/jimmunol.174.7.4345. PMID 15778399
- [Background] Serhan CN, Clish CB, Brannon J, Colgan SP, Chiang N, Gronert K. Novel functional sets of lipid-derived mediators with antiinflammatory actions generated from omega-3 fatty acids via cyclooxygenase 2-nonsteroidal antiinflammatory drugs and transcellular processing. J Exp Med. 2000 Oct 16;192(8):1197-204. doi: 10.1084/jem.192.8.1197. PMID 11034610
- [Background] Grenon SM, Aguado-Zuniga J, Hatton JP, Owens CD, Conte MS, Hughes-Fulford M. Effects of fatty acids on endothelial cells: inflammation and monocyte adhesion. J Surg Res. 2012 Sep;177(1):e35-43. doi: 10.1016/j.jss.2012.04.010. Epub 2012 Apr 27. PMID 22572621
- [Background] Yang R, Chiang N, Oh SF, Serhan CN. Metabolomics-lipidomics of eicosanoids and docosanoids generated by phagocytes. Curr Protoc Immunol. 2011 Nov;Chapter 14:Unit 14.26. doi: 10.1002/0471142735.im1426s95. PMID 22048801
- [Background] Tang Y, Zhang MJ, Hellmann J, Kosuri M, Bhatnagar A, Spite M. Proresolution therapy for the treatment of delayed healing of diabetic wounds. Diabetes. 2013 Feb;62(2):618-27. doi: 10.2337/db12-0684. Epub 2012 Oct 5. PMID 23043160
- [Background] Harris WS. The omega-3 index as a risk factor for coronary heart disease. Am J Clin Nutr. 2008 Jun;87(6):1997S-2002S. doi: 10.1093/ajcn/87.6.1997S. PMID 18541601
- [Background] Freidlin B, Korn EL, George SL. Data monitoring committees and interim monitoring guidelines. Control Clin Trials. 1999 Oct;20(5):395-407. doi: 10.1016/s0197-2456(99)00017-3. PMID 10503800
- [Background] Whitehead J. Monitoring and evaluating clinical trials data. Intensive Care Med. 2000;26 Suppl 1:S84-8. doi: 10.1007/s001340051123. PMID 10786963
- [Background] Morse MA, Califf RM, Sugarman J. Monitoring and ensuring safety during clinical research. JAMA. 2001 Mar 7;285(9):1201-5. doi: 10.1001/jama.285.9.1201. PMID 11231751